CLINICAL TRIAL: NCT03637868
Title: A Phase II Study of Eribulin in Brain Metastases From HER2-negative Breast Cancer Pre-treated With Anthracyclines and Taxanes
Brief Title: Eribulin in Brain Metastases From HER2-negative Breast Cancer
Acronym: ERIBRAIN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no enrollment
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERIBRAIN-IPC 2017-014; 2018-001027-40 (EudraCT Number)
Record Dates: First submitted 2018-08-06; First posted 2018-08-20 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-negative breast cancer; brain metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — eribulin

STUDY DESIGN:
Intervention Model Description: Prospective, national, multicenter, open-label, uncontrolled, multi-cohort phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eribulin (Experimental): eribulin 1.4 mg/m² administered intravenously between 6 and 7 cycles.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — Patients will receive eribulin 1.4 mg/m² administered intravenously over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle.

SUMMARY:
To evaluate the efficacy of eribulin for treatment of HER2-negative breast cancer brain metastases (BCBM)

DETAILED DESCRIPTION:
This study will explore eribulin in three specific cohorts of patients with HER2-negative metastatic breast cancer harboring BCBM, pretreated with anthracyclines and taxanes:

* Cohort A = Newly diagnosed, untreated BCBM, not candidate to initial surgery or stereotactic radiosurgery (SRS) and with pauci-symptomatic disease not requiring immediate whole-brain radiation therapy (WBRT)
* Cohort B = BCBM pretreated with SRS and/or surgery alone, without WBRT, and not requiring immediate WBRT
* Cohort C = BCBM pretreated with WBRT

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Life expectancy of 3 months or longer.
3. ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2.
4. HER2-negative (IHC 0/1+ or 2+ and in situ hybridization negative) metastatic breast cancer
5. Locally advanced or metastatic breast cancer that have progressed after at least one chemotherapeutic regimen for advanced disease. Prior therapy should have included an anthracycline and a taxane in either the adjuvant or metastatic setting unless patients were not suitable for these treatments. (no limit to the number of previous lines of therapy, no need for extracranial disease)
6. At least 2 weeks washout period post chemotherapy, targeted or biologic therapy, or radiation therapy is required prior to study entry
7. Patient with untreated CNS disease or previous SRS/surgery without WBRT (cohorts A and B)

   * At least 1 measurable CNS lesion ≥ 10 mm on T1-weighted gadolinium-enhanced MRI, OR
   * At least one CNS tumor measuring 5-9 mm in longest diameter, plus one or two additional CNS tumors measuring ≥ 3 mm in longest diameter, for which the sum of the longest diameters is ≥ 10 mm.
8. Patient with progressive disease harboring brain metastases after previous WBRT (cohort C)

   * At least 1 measurable CNS lesion ≥ 10 mm on T1-weighted gadolinium-enhanced MRI, OR
   * At least one CNS tumor measuring 5-9 mm in longest diameter, plus one or two additional CNS tumors measuring ≥ 3 mm in longest diameter, for which the sum of the longest diameters is ≥ 10 mm.
9. Adequate organ function as evidenced by:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10e9/L without granulocyte-colony-stimulating factor G-CSF (filgrastim, pegfilgrastim, or equivalent) support within 7 days
   * Hemoglobin (Hgb) ≥ 9.0 g/dL (90 g/L) without blood transfusion within 7 days
   * Platelet count ≥ 100 x 10e9/L without platelet transfusion within 7 days
   * Bilirubin ≤ 1.5 X upper limit of normal (ULN), except for patients with documented history of Gilbert's disease who may have DIRECT bilirubin ≤ 1.5 X ULN
   * Alanine aminotransferase (ALT) ≤ 2.5 X ULN, except ≤ 5 X ULN for patients with liver metastases
   * Aspartate aminotransferase (AST) ≤ 2.5 X ULN, except ≤ 5 X ULN for patients with liver metastases
   * Serum creatinine ≤ 1.5 X ULN; or calculated creatinine clearance ≥ 50 mL/min (using MDRD formula), or measured creatinine clearance ≥ 50 mL/min

Exclusion Criteria:

1. Prior therapy with eribulin.
2. Patients should not have had major surgery or radiotherapy (therapeutic and/or palliative) within 14 days prior to initiation of study treatment, including CNS-directed radiation therapy. (Minor procedures, such as tumor biopsy, thoracentesis, or intravenous catheter placement are allowed with no waiting period)
3. Patients may not have the following co morbid disease or concurrent illness:

   * Known cirrhosis, defined as Child Pugh class A or higher liver disease
   * Other active malignancy, except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder)
   * Any other severe/uncontrolled inter current illness or significant co morbid conditions that in the opinion of the investigator would impair study participation or cooperation
   * Patients with the presence of an active infection, abscess or fistula
   * Known leptomeningeal disease or CNS midline shifts.
   * Any evidence of severe or uncontrolled systemic disease such as clinically significant cardiovascular, pulmonary, hepatic, renal or metabolic disease.
   * Severe conduction abnormality including significant corrected QT interval QTc prolongation >450ms.
   * Patients with grade 3/4 peripheral neuropathy.
4. Patient candidate to SRS and or surgical resection
5. Major clinical symptoms requiring immediate WBRT as defined by "local tumor board"
6. Increase in corticosteroid dose in the week prior to baseline brain MRI
7. Patients with pacemaker or implantable cardioverter-defibrillator devices incompatible with MRI assessment.
8. Contraindication to Gadolinium infusion.
9. Treatment ongoing with other chemotherapy, hormonal therapy, immunotherapy, other investigational agents, or biologic agents for the treatment of cancer except bisphosphonates or denosumab.
10. Pregnant or breast-feeding patients
11. Women of child-bearing potential without effective contraception method.
12. Patient unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of eribulin for treatment of HER2-negative BCBM | from inclusion until 30 days after completion of treatment
  By estimating central nervous system (CNS) objective response rate per RANO-BM criteria. CNS objective response rate will be defined as the rate of patients with a partial response or a complete response as defined by RANO-BM criteria (Lin et al. 2015)

SECONDARY OUTCOMES:
Safety of Eribulin in this population | from Eribulin initiation until 30 days after completion of treatment
  Toxicity will be evaluated before every chemotherapy infusion according to NCI CTCAE v5.0 criteria. All treatment-related adverse events will be collected. The rate of grade 3 to 5 adverse events will be analyzed
Time to WBRT (cohort A and B) | from Eribulin initiation to the time of the first dose of whole brain radiation therapy - up to 28 months
  Time to WBRT will be defined as the time from Eribulin initiation to WBRT start
CNS progression-free survival | from Eribulin initiation until the date of first documented CNS disease progression or date of death from any cause - up to 28 months
  CNS progression-free survival will be defined as the time from Eribulin initiation to CNS disease progression according to RANO-BM criteria or death from any cause
Overall survival | from Eribulin initiation to death
  Overall survival will be defined as the time from Eribulin initiation to death from any cause
Change in cognitive function | From Eribulin initiation up to 7 days after study treatment discontinuation
  Cognitive function will be evaluated by self-report Fact-Cog v3.0 questionnaires (French validated version;(Joly et al. 2012)) that will have to be filled every two cycles (before every day 1 infusion)
Quality of life measured by Functional Assessment of Cancer Therapy-Brain Metastasis | From Eribulin initiation up to 7 days after study treatment discontinuation
  Quality of life will be measured by Functional Assessment of Cancer Therapy-Brain Metastasis (FACT-Br v4.0, (Thavarajah et al. 2014)) questionnaire. This questionnaire will be filled every two cycles

OTHER OUTCOMES:
Progression-free survival for non-CNS disease | from Eribulin initiation until the date of first documented extra-cranial disease progression or date of death from any cause - up to 28 months
  Extracranial progression-free survival will be defined as the time from Eribulin initiation to disease progression according to RECIST 1.1 criteria (Schwartz et al. 2016) or death from any cause. Thoracic and abdominal CT-scans will be performed as recommended in each participating center (usually every 6 weeks) to assess non CNS disease (extracranial PFS, non-CNS response rate, and clinical benefit). Non-CNS disease will be evaluated according to investigator assessment.
Bi-compartmental progression-free survival (PFS) | from Eribulin initiation until the date of first documented progression or date of death from any cause - up to 28 months
  Bi-compartmental PFS will be defined as the time from Eribulin initiation to CNS disease progression according to RANO-BM criteria or non-CNS disease progression according to RECIST 1.1 criteria or death from any cause
Overall response rate for extra-CNS disease | from Eribulin initiation until 30 days after completion of treatment
  The overall response rate for non-CNS disease will be defined as the rate of patients with a partial response or a complete response according to RECIST 1.1 criteria
Clinical benefit for both CNS and extra-CNS disease | partial response or complete response or disease stabilization > 6 months
  The clinical benefit rate will be defined as the rate of patients with a partial response or a complete response or disease stabilization > 6 months. Clinical benefit will be assessed for both CNS (using RANO-BM criteria) and non-CNS disease (using RECIST 1.1 criteria), separately
Eribulin efficacy according to hormone receptors expression | from Eribulin initiation until 30 days after completion of treatment
  CNS objective response rates will be assessed according to hormone receptors expression (positive vs negative). A case will be defined as hormone receptors negative if both estrogen receptor and progesterone receptor expression are expressed by less than 10% of tumor cells
Efficacy comparison between patients with and without non-CNS disease | from Eribulin initiation until 30 days after completion of treatment
  CNS objective response rates will be assessed according the presence of non-CNS disease ('CNS only' vs 'not CNS only').

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Sabatier, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (7):
- France (7):
  - Institut de Cancerologie de L'Ouest - Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - CHU Besançon, Besançon
  - Institut Paoli-Calmettes, Marseille
  - Institut Du Cancer de Montpellier, Montpellier
  - Institut De Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancerologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arslan C, Dizdar O, Altundag K. Chemotherapy and biological treatment options in breast cancer patients with brain metastasis: an update. Expert Opin Pharmacother. 2014 Aug;15(12):1643-58. doi: 10.1517/14656566.2014.929664. PMID 25032884
- [Background] Bart J, Nagengast WB, Coppes RP, Wegman TD, van der Graaf WT, Groen HJ, Vaalburg W, de Vries EG, Hendrikse NH. Irradiation of rat brain reduces P-glycoprotein expression and function. Br J Cancer. 2007 Aug 6;97(3):322-6. doi: 10.1038/sj.bjc.6603864. Epub 2007 Jul 3. PMID 17609666
- [Background] Bartsch R, Fromm S, Rudas M, Wenzel C, Harbauer S, Roessler K, Kitz K, Steger GG, Weitmann HD, Poetter R, Zielinski CC, Dieckmann K. Intensified local treatment and systemic therapy significantly increase survival in patients with brain metastases from advanced breast cancer - a retrospective analysis. Radiother Oncol. 2006 Sep;80(3):313-7. doi: 10.1016/j.radonc.2006.08.001. Epub 2006 Sep 7. PMID 16959347
- [Background] Chang AY, Ying XX. Brain Metastases from Breast Cancer and Response to Treatment with Eribulin: A Case Series. Breast Cancer (Auckl). 2015 May 24;9:19-24. doi: 10.4137/BCBCR.S21176. eCollection 2015. PMID 26052228
- [Background] Cortes J, O'Shaughnessy J, Loesch D, Blum JL, Vahdat LT, Petrakova K, Chollet P, Manikas A, Dieras V, Delozier T, Vladimirov V, Cardoso F, Koh H, Bougnoux P, Dutcus CE, Seegobin S, Mir D, Meneses N, Wanders J, Twelves C; EMBRACE (Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389) investigators. Eribulin monotherapy versus treatment of physician's choice in patients with metastatic breast cancer (EMBRACE): a phase 3 open-label randomised study. Lancet. 2011 Mar 12;377(9769):914-23. doi: 10.1016/S0140-6736(11)60070-6. Epub 2011 Mar 2. PMID 21376385
- [Background] Jimeno A. Eribulin: rediscovering tubulin as an anticancer target. Clin Cancer Res. 2009 Jun 15;15(12):3903-5. doi: 10.1158/1078-0432.CCR-09-1023. Epub 2009 Jun 9. PMID 19509144
- [Background] Joly F, Lange M, Rigal O, Correia H, Giffard B, Beaumont JL, Clisant S, Wagner L. French version of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) version 3. Support Care Cancer. 2012 Dec;20(12):3297-305. doi: 10.1007/s00520-012-1439-2. Epub 2012 May 2. PMID 22549504
- [Background] Jordan MA, Kamath K, Manna T, Okouneva T, Miller HP, Davis C, Littlefield BA, Wilson L. The primary antimitotic mechanism of action of the synthetic halichondrin E7389 is suppression of microtubule growth. Mol Cancer Ther. 2005 Jul;4(7):1086-95. doi: 10.1158/1535-7163.MCT-04-0345. PMID 16020666
- [Background] Kaufman PA, Awada A, Twelves C, Yelle L, Perez EA, Velikova G, Olivo MS, He Y, Dutcus CE, Cortes J. Phase III open-label randomized study of eribulin mesylate versus capecitabine in patients with locally advanced or metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2015 Feb 20;33(6):594-601. doi: 10.1200/JCO.2013.52.4892. Epub 2015 Jan 20. PMID 25605862
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Barboriak DP, Baumert BG, Bendszus M, Brown PD, Camidge DR, Chang SM, Dancey J, de Vries EG, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Response assessment criteria for brain metastases: proposal from the RANO group. Lancet Oncol. 2015 Jun;16(6):e270-8. doi: 10.1016/S1470-2045(15)70057-4. Epub 2015 May 27. PMID 26065612
- [Background] Lu J, Steeg PS, Price JE, Krishnamurthy S, Mani SA, Reuben J, Cristofanilli M, Dontu G, Bidaut L, Valero V, Hortobagyi GN, Yu D. Breast cancer metastasis: challenges and opportunities. Cancer Res. 2009 Jun 15;69(12):4951-3. doi: 10.1158/0008-5472.CAN-09-0099. Epub 2009 May 26. No abstract available. PMID 19470768
- [Background] Matsuoka H, Tsurutani J, Tanizaki J, Iwasa T, Komoike Y, Koyama A, Nakagawa K. Regression of brain metastases from breast cancer with eribulin: a case report. BMC Res Notes. 2013 Dec 18;6:541. doi: 10.1186/1756-0500-6-541. PMID 24350786
- [Background] Narayan S, Carlson EM, Cheng H, Condon K, Du H, Eckley S, Hu Y, Jiang Y, Kumar V, Lewis BM, Saxton P, Schuck E, Seletsky BM, Tendyke K, Zhang H, Zheng W, Littlefield BA, Towle MJ, Yu MJ. Novel second generation analogs of eribulin. Part III: Blood-brain barrier permeability and in vivo activity in a brain tumor model. Bioorg Med Chem Lett. 2011 Mar 15;21(6):1639-43. doi: 10.1016/j.bmcl.2011.01.096. Epub 2011 Jan 26. PMID 21324687
- [Background] Pivot X, Marme F, Koenigsberg R, Guo M, Berrak E, Wolfer A. Pooled analyses of eribulin in metastatic breast cancer patients with at least one prior chemotherapy. Ann Oncol. 2016 Aug;27(8):1525-31. doi: 10.1093/annonc/mdw203. Epub 2016 May 13. PMID 27177860
- [Background] Qin DX, Zheng R, Tang J, Li JX, Hu YH. Influence of radiation on the blood-brain barrier and optimum time of chemotherapy. Int J Radiat Oncol Biol Phys. 1990 Dec;19(6):1507-10. doi: 10.1016/0360-3016(90)90364-p. PMID 2262373
- [Background] Schwartz LH, Litiere S, de Vries E, Ford R, Gwyther S, Mandrekar S, Shankar L, Bogaerts J, Chen A, Dancey J, Hayes W, Hodi FS, Hoekstra OS, Huang EP, Lin N, Liu Y, Therasse P, Wolchok JD, Seymour L. RECIST 1.1-Update and clarification: From the RECIST committee. Eur J Cancer. 2016 Jul;62:132-7. doi: 10.1016/j.ejca.2016.03.081. Epub 2016 May 14. PMID 27189322
- [Background] Thavarajah N, Bedard G, Zhang L, Cella D, Beaumont JL, Tsao M, Barnes E, Danjoux C, Sahgal A, Soliman H, Chow E. Psychometric validation of the functional assessment of cancer therapy--brain (FACT-Br) for assessing quality of life in patients with brain metastases. Support Care Cancer. 2014 Apr;22(4):1017-28. doi: 10.1007/s00520-013-2060-8. Epub 2013 Nov 28. PMID 24287508
- [Background] Toth K, Vaughan MM, Peress NS, Slocum HK, Rustum YM. MDR1 P-glycoprotein is expressed by endothelial cells of newly formed capillaries in human gliomas but is not expressed in the neovasculature of other primary tumors. Am J Pathol. 1996 Sep;149(3):853-8. PMID 8780389
- [Background] Zhang RD, Price JE, Fujimaki T, Bucana CD, Fidler IJ. Differential permeability of the blood-brain barrier in experimental brain metastases produced by human neoplasms implanted into nude mice. Am J Pathol. 1992 Nov;141(5):1115-24. PMID 1443046